CLINICAL TRIAL: NCT05669625
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Live Attenuated Varicella Vaccine in Healthy People
Brief Title: A Phase III Clinical Trial to Evaluate the Efficacy and Safety of the Live Attenuated Varicella Vaccine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Jiangsu Province Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CNBG-BIBP-VZV-07
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Varicella
Keywords: vaccine efficacy; varicella vaccine; safety; immunogenicity
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Single subcutaneous injection of the investigational vaccine (0.5 ml)
  Interventions: Biological: Investigational live attenuated varicella vaccine
- Placebo Group (Placebo Comparator): Single subcutaneous injection of the investigational placebo (0.5 ml)
  Interventions: Biological: Placebo of live attenuated varicella vaccine

INTERVENTIONS:
Biological: Investigational live attenuated varicella vaccine — 0.5 ml/vial
  Arms: Experimental Group
Biological: Placebo of live attenuated varicella vaccine — 0.5 ml/vial
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety and immunogenicity of a live attenuated varicella vaccine manufactured by Beijing Institute of Biological Products Co., Ltd in healthy children.

DETAILED DESCRIPTION:
This trial is aim to evaluate the efficacy, safety and immunogenicity of a live attenuated varicella vaccine manufactured by Beijing Institute of Biological Products Co., Ltd in healthy children aged 1-12 years old.

This study will be conducted in two stage. the stage 1 adopts an open design, and 20 subjects aged 18~59 and 13~17 years old (18~59 years old→ 13~17 years old, sequentially enrolled) are enrolled, and 1 dose of the trial vaccine is administered to explore safety.

The stage 2 adopts a randomized, blinded, placebo-controlled design, 12400 healthy participants aged 1-12 years old will be randomly assigned into experimental group or control group with the ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 13 - 59 years old for Stage 1, 1-12 years old for Stage 2, and be able to provide legal identification ;
* Subject and/or guardian has the ability to understand study requirements and processes, consent to participate in clinical trials, and sign informed consent forms;
* Consent to use effective contraception during study participation, no pregnancy and no family planning (for women of childbearing potential or their spouses);
* Axillary temperature ≤ 37.0 °C on the day of enrollment;

Exclusion Criteria:

* Has received any varicella vaccine before ( Not applicable to Stage 1）;
* Has history of varicella or herpes zoster infection, or contact with varicella/shingles patients or suspected varicella/shingles patients within 30 days before enrollment ( Not applicable to Stage 1）;
* Currently using salicylates (including salicylic acid, aspirin, diflunisalin, p-aminosalicylate (sodium), dicalicylate, benoxate, etc.), or plan to use it for a long time during the study；
* Have had febrile illness (axillary temperature ≥ 38.5 °C) or used antipyretic, analgesic, anti-allergic drugs (such as acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) 3 days before vaccination；
* Have a history of allergy to vaccine components and excipients or severe drug allergy, such as anaphylactic shock, allergic laryngeal edema, Henoch-Schönlein purpura, thrombocytopenic purpura, local allergic necrosis (Arthus) reaction, severe urticaria, etc；
* Have a history of epilepsy, convulsions or convulsions, and have a family history of severe neurological disease or psychosis
* Immunocompromised or diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune diseases；
* With severe congenital malformations, hereditary diseases, serious cardiovascular diseases, serious liver/kidney diseases, complicated diabetes, malignant tumors, and severe malnutrition
* Immunosuppressant therapy, such as long-term oral or injectable glucocorticoid therapy (≥ 14 days, dose ≥2 mg/kg/day or ≥20 mg/day or equivalent to prednisone), within 3 months prior to enrollment or planned within 30 days of vaccination, but topical medications (e.g., ointments, eye drops, inhalers, or nasal sprays) are not restricted
* Have received blood/blood-related products or immunoglobulins 3 months prior to vaccination, or plan to use such products 30 days after vaccination；
* Have received a live attenuated vaccine within 30 days prior to the trial vaccine, or any vaccine within 14 days prior to vaccination;
* Asplenectomy or splenectomy due to any condition (e.g. splenectomy);
* Those with a history of thrombocytopenia or other coagulation disorders, which may cause contraindications to subcutaneous injection;
* Suffering from various infectious, purulent or allergic skin diseases;
* Are participating in other investigational or unregistered clinical trials of products (drugs, vaccines or devices, etc.), or have plans to participate in other clinical trials before the end of this clinical trial;
* Has any other factors that are not suitable for participation in the clinical trial in the judgment of the investigator

Ages: 1 Year to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12440 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-04-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
The incidences of varicella in each group | number of cases reported 30 days after vaccination
  The first 24 cases of varicella occurred 30 days after injection will be collected
The efficacy of the live attenuated varicella vaccine | number of cases reported 30 days after vaccination
  The vaccine efficacy will be calculated based on the reported cases occurred 30 days after vaccination

SECONDARY OUTCOMES:
The vaccine efficacy against laboratory-confirmed cases of moderate and severe varicella | number of cases reported 30 days after vaccination
  The vaccine efficacy will be calculated based on the reported cases occurred 30 days after vaccination
The vaccine efficacy against clinical-confirmed cases | number of cases reported 30 days after vaccination
  calculated based on the reported cases occurred 30 days after vaccination
The incidences of adverse events (AEs) | within 30 days after vaccination
  AEs occurred within 30 days after injection will be collected
The incidences of serious adverse events (SAEs) | at least 6 months after vaccination
  SAEs occurred within 6 months after vaccination will be collected
The geometric mean titer (GMT) in the immunogenicity subgroup | 30 days after vaccination
  Geometric mean titer (GMT) will be measured before and 30 days after vaccination
The seroconversion rate of the immunogenicity subgroup | 30 days after vaccination
  The seroconversion rate will be calculated before and 30 days after vaccination
The geometric mean fold increase (GMI) of the immunogenicity subgroup | 30 days after vaccination
  Geometric mean fold increase (GMI) of the immunogenicity group will be calculated based on the geometric mean titer
The immune persistence of the immunogenicity subgroup | 1 year, 2 years, and 3 years after vaccination
  Geometric mean titer (GMT) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Principal Investigator — Jiangsu Province Centers for Disease Control and Prevention
Locations (13):
- China (13):
  - Sinan County Center for Disease Control and Prevention, Tongren, Guizhou
  - Songtao Miao Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou
  - Yuping Dong Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou
  - Qi County Center for Disease Control and Prevention, Hebi, Henan
  - Wuzhi County Center for Disease Control and Prevention, Jiaozuo, Henan
  - Wuyang County Center for Disease Control and Prevention, Luohe, Henan
  - Pei County Center for Disease Control and Prevention, Xuzhou, Jiangsu
  - Huaiyin District Center for Disease Control and Prevention, Xuzhou, Jiangsu
  - Mianyang Anzhou District Center for Disease Control and Prevention, Mianyang, Sichuan
  - Southern County Center for Disease Control and Prevention, Nanchong, Sichuan
  - Neijiang City Center for Disease Control and Prevention, Neijiang, Sichuan
  - Lancang Lahu Autonomous County Center for Disease Control and Prevention, Pu'er, Yunnan
  - Yanshan County Center for Disease Control and Prevention, Wenshan, Yunnan

IPD SHARING:
Plan to Share IPD: No